CLINICAL TRIAL: NCT02499263
Title: A Prospective Multicenter Study to Observe the Effectiveness on Ulcerative Colitis and Predictive Factors of Clinical Response in Korean Patients Treated With Adalimumab (EUREKA Study)
Brief Title: A Prospective Non-interventional Multicenter Study to Evaluate the Effectiveness of Adalimumab in Korean Patients With Ulcerative Colitis (UC) and Identify Potential Predictors of Clinical Response in Routine Clinical Practice
Acronym: EUREKA
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-346
Record Dates: First submitted 2015-07-01; First posted 2015-07-16 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Ulcerative Colitis
Keywords: Adalimumab trough level; Fecal Calprotectin; Fecal microbiota
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fecal samples : Fecal calprotectin and the composition of Fecal microbiota. Blood samples : Trough level of adalimumab & Antibodies against adalimumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Ulcerative Colitis (UC): Adalimumab 160 mg at week 0, 80 mg at week 2, and then 40 mg every other week per the Korean label in participants with active moderate-to-severe UC.

SUMMARY:
This is a prospective, single country, multi-center study in participants with ulcerative colitis (UC) treated with adalimumab. Up to 147 participants are enrolled at approximately 20 sites. The baseline assessment is performed prior to the first dose of adalimumab (Visit 1). Study visits are conducted at weeks 8, 16, 24, 32, 40, 48 and 56 after baseline in accordance with clinical practice. All participants will have one Follow-up for safety approximately 70 days after the last dose of adalimumab.

DETAILED DESCRIPTION:
This is a prospective, single-country, multi-center study in UC patients treated with adalimumab. The prescription of adalimumab is at the discretion of the physician in accordance with clinical practice and label, is made independently from this study, and preceded the decision to offer the patient the opportunity to participate in this study.

Up to 147 subjects are planned to be enrolled at approximately 20 sites. The baseline assessment is performed prior to the first dose of adalimumab (Visit 1). Participants are administered adalimumab 160 mg at Week 0, 80 mg at Week 2, and then 40 mg every other week per the Korean label. Study visits are conducted at Weeks 8, 16, 24, 32, 40, 48 and 56 after baseline in accordance with clinical practice. All participants had one Follow-up for safety approximately 70 days after the last dose of adalimumab.

Clinical response is assessed at Week 8, and participants with clinical response at Week 8 can continue on adalimumab treatment as per Korean reimbursement guidelines. Clinical response is defined as a decrease from baseline in the total Mayo score by at least 3 points and at least 30% with an accompanying decrease in rectal bleeding subscore of at least 1 point or absolute rectal bleeding sub-score of 0 or 1.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be an adult ≥19 years
* Participant with active moderate to severe ulcerative colitis with Mayo score of ≥ 6 points and endoscopic sub-score of ≥ 2 points despite treatment with corticosteroids and/or immunosuppressants.
* Participant must have tuberculosis (TB) Screening Assessment in accordance Korean reimbursement guidelines.
* Participants who had started on adalimumab treatment in normal clinical practice setting by their physician.
* Participant must provide written authorization form to use personal and/or health data prior to the entry into the study.

Exclusion Criteria:

* Female participants who are pregnant or breast feeding
* Participant with any contraindication to adalimumab
* Participant that is participating in other clinical trials

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with moderate to severe ulcerative colitis (UC) receiving adalimumab per the Korean label.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (19):
- South Korea (19):
  - Kyungpook National Univ Hosp /ID# 153133, Daegu, Daegu Gwang Yeogsi
  - St. Vincent's Hospital /ID# 138455, Suwon, Gyeonggido
  - Ajou University Hospital /ID# 138457, Suwon, Gyeonggido
  - Inje University Busan Paik Hospital /ID# 138451, Pusan, Gyeongsangbuk-do
  - Inha University Hospital /ID# 150176, Junggu, Incheon Gwang Yeogsi
  - Chonnam National University Hospital /ID# 138450, Gwangju, Jeonranamdo
  - Kyung Hee University Medical Center /ID# 138453, Dongdaemun-gu, Seoul Teugbyeolsi
  - Kangbuk Samsung Hospital /ID# 150175, Jongno-Gu, Seoul Teugbyeolsi
  - Severance Hospital /ID# 138456, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 138449, Seoul, Seoul Teugbyeolsi
  - SMG-SNU Boramae Medical Center /ID# 138448, Seoul, Seoul Teugbyeolsi
  - Keimyung Univ Dongsan medical /ID# 138447, Daegu
  - Daejeon St. Mary's Hospital /ID# 138445, Daejeon
  - Chosun University Hospital /ID# 138454, Gwangju
  - Korea University Anam Hospital /ID# 138446, Seoul
  - Seoul National University Hospital /ID# 138443, Seoul
  - Ewha Womans University Mokdong /ID# 138444, Seoul
  - Inje University Seoul Paik Hos /ID# 138452, Seoul
  - Chung-Ang University Med. Ctr. /ID# 138441, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Regarding Medicine Information — http://rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 150 participants enrolled; 4 were not treated and hence 146 were included in the intent to treat (ITT) set.
Groups:
- Adalimumab: Adalimumab 160 mg at week 0, 80 mg at week 2, and then 40 mg every other week per the Korean label.
Period: Overall Study
Arm/Group | Adalimumab
Started | 146
Completed | 84
Not Completed | 62
Not completed — Lost to Follow-up | 9
Not completed — Participant's withdrawal of consent | 4
Not completed — Lack of Efficacy | 22
Not completed — investigator's judgment | 12
Not completed — Adverse Events/Serious Adverse Events | 11
Not completed — Participant's decision | 3
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Population: ITT set: all participants intended to be treated with adalimumab. At week 8, all participants who had received adalimumab treatment at least once were included and at week 56, all participants who had clinical response at week 8 were included.
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.96 (14.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 96
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Week 8 Responders With Durable Clinical Response at Week 56
Description: Durable clinical response was defined as reduction in complete Full Mayo score of ≥3 points and ≥30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point at both Week 8 and 56. Clinical response was defined as reduction in complete full Mayo score of ≥3 points and ≥30% from Baseline (Week 0) with decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point at Week 8. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and physician's global assessment [PGA]), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Week 56
Population: ITT set: all participants that were intended to be treated with adalimumab. At Week 8, all participants who had received adalimumab treatment at least once were included and at Week 56, all participants who had clinical response at Week 8 were included. A participant was a Week 8 responder if they had a clinical response at Week 8.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 76
percentage of participants | 53.95 [42.13 to 65.45]

2. Primary Outcome: Percentage of Participants With Clinical Response at Week 8
Description: Clinical response was defined as reduction in complete full Mayo score of ≥3 points and ≥30% from Baseline (Week 0) with decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point at week 8. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and PGA), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Week 8
Population: ITT set: all participants that were intended to be treated with adalimumab. At Week 8, all participants who had received adalimumab treatment at least once were included and at Week 56, all participants who had clinical response at Week 8 were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
percentage of participants | 52.05 [43.64 to 60.38]

3. Primary Outcome: Percentage of Participants With Clinical Response at Week 24
Description: Clinical response was defined as reduction in complete full Mayo score of ≥3 points and ≥30% from Baseline (Week 0) with decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point at Week 24. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and PGA), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Week 24
Population: ITT set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
percentage of participants | 54.11 [45.67 to 62.38]

4. Primary Outcome: Percentage of Participants With Clinical Response at Week 56
Description: Clinical response was defined as reduction in complete full Mayo score of ≥3 points and ≥30% from Baseline (Week 0) with decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point at Week 56. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and PGA), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Week 56
Population: ITT set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
percentage of participants | 37.67 [29.79 to 46.06]

5. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 8
Description: Clinical remission was defined as the full Mayo score ≤2 points, with no individual sub-score exceeding 1 point at Week 8. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and PGA), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Week 8
Population: ITT set
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
percentage of participants | 23.97

6. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 56
Description: Clinical remission was defined as the full Mayo score ≤2 points, with no individual sub-score exceeding 1 point at Week 56. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and PGA), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Week 56
Population: ITT set
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
percentage of participants | 21.92

7. Secondary Outcome: Percentage of Participants Who Were Week 8 Responders With Clinical Remission at Week 8
Description: Clinical remission was defined as the full Mayo score ≤2 points, with no individual sub-score exceeding 1 point at Week 8. Clinical response was defined as reduction in complete full Mayo score of ≥ 3 points and ≥ 30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥ 1 point or absolute rectal bleeding subscore of ≤ 1 point at Week 8. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and PGA), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Week 8
Population: ITT set. A participant was a Week 8 responder if they had a clinical response at Week 8.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
percentage of participants | 23.97

8. Secondary Outcome: Percentage of Participants Who Were Week 8 Responders With Clinical Remission at Week 56
Description: Clinical remission was defined as the full Mayo score ≤2 points, with no individual sub-score exceeding 1 point at Week 56. Clinical response was defined as reduction in complete full Mayo score of ≥ 3 points and ≥ 30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥ 1 point or absolute rectal bleeding subscore of ≤ 1 point at Week 8. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and PGA), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Week 56
Population: ITT set. A participant was a Week 8 responder if they had a clinical response at Week 8.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 76
percentage of participants | 35.53

9. Secondary Outcome: Percentage of Participants With Steroid-free Remission at Week 8
Description: Steroid free remission was defined as participants who were in remission without the use of systemic steroids from Visit 1 (Baseline) prior to assessment.
Time Frame: Week 8
Population: ITT set
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
percentage of participants | 12.33

10. Secondary Outcome: Percentage of Participants With Steroid-free Remission at Week 56
Description: Steroid free remission was defined as participants who were in remission without the use of systemic steroids within the past 12 weeks prior to assessment.
Time Frame: Week 56
Population: ITT set
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
percentage of participants | 21.23

11. Secondary Outcome: Percentage of Participants Who Were Week 8 Responders With Steroid-free Remission at Week 8
Description: Steroid-free remission was defined as participants who were in remission without the use of systemic steroids within the past 12 weeks prior to assessment. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. Clinical response was defined as reduction in complete full Mayo score of ≥ 3 points and ≥ 30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥ 1 point or absolute rectal bleeding subscore of ≤ 1 point at Week 8. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and PGA), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Week 8
Population: ITT set. A participant was a Week 8 responder if they had a clinical response at Week 8.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
percentage of participants | 12.33

12. Secondary Outcome: Percentage of Participants Who Were Week 8 Responders With Steroid-free Remission at Week 56
Description: Steroid free remission was defined as participants who were in remission without the use of systemic steroids within the past 12 weeks prior to assessment. Clinical response was defined as reduction in complete full Mayo score of ≥ 3 points and ≥ 30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥ 1 point or absolute rectal bleeding subscore of ≤ 1 point at Week 8. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and PGA), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Week 56
Population: ITT set. A participant was a Week 8 responder if they had a clinical response at Week 8.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 76
percentage of participants | 34.21

13. Secondary Outcome: Percentage of Participants With Steroid-free Response at Week 8
Description: Steroid-free response was defined as participants who were in clinical response without the use of systemic steroids within the past 8 weeks prior to assessment. Clinical response was defined as reduction in complete full Mayo score of ≥ 3 points and ≥ 30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥ 1 point or absolute rectal bleeding subscore of ≤ 1 point at Week 8. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and PGA), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Week 8
Population: ITT set.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
percentage of participants | 30.82

14. Secondary Outcome: Percentage of Participants With Steroid-free Response at Week 56
Description: as for outcome 13
Time Frame: Week 56
Population: ITT set.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
percentage of participants | 36.30

15. Secondary Outcome: Percentage of Participants Who Were Week 8 Responders With Steroid-free Response at Week 8
Description: Steroid free response was defined as participants who were in clinical response without the use of systemic steroids within the past 8 weeks prior to assessment (in Week 8 clinical responders).Clinical response was defined as reduction in complete full Mayo score of ≥ 3 points and ≥ 30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥ 1 point or absolute rectal bleeding subscore of ≤ 1 point at Week 8. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and PGA), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Week 8
Population: ITT set. A participant was a Week 8 responder if they had a clinical response at Week 8.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
percentage of participants | 30.82

16. Secondary Outcome: Percentage of Participants Who Were Week 8 Responders With Steroid-free Response at Week 56
Description: Steroid free response was defined as participants who were in clinical response without the use of systemic steroids within the past 12 weeks prior to assessment (in Week 8 clinical responders). A participant was a Week 8 responder if they had a clinical response at Week 8. Clinical response was defined as reduction in complete full Mayo score of ≥ 3 points and ≥ 30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥ 1 point or absolute rectal bleeding subscore of ≤ 1 point at Week 8. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and PGA), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Week 56
Population: ITT set. A participant was a Week 8 responder if they had a clinical response at Week 8.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 76
percentage of participants | 51.32

17. Secondary Outcome: Percentage of Participants With Mucosal Healing at Week 8
Description: Mucosal healing was defined as an endoscopy sub-score of 0 or 1 at week 8. Endoscopic findings were scored on a scale from 0 to 3 as follows:
  0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern, mild friability); 2 = Moderate disease (marked erythema, lack of vascular pattern, friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration). The higher the score, the more severe the disease.
Time Frame: Week 8
Population: ITT set
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
percentage of participants | 39.04

18. Secondary Outcome: Percentage of Participants With Mucosal Healing at Week 56
Description: Mucosal healing was defined as an endoscopy sub-score of 0 or 1 at Week 56. Endoscopic findings were scored on a scale from 0 to 3 as follows:
  0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern, mild friability); 2 = Moderate disease (marked erythema, lack of vascular pattern, friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration). The higher the score, the more severe the disease.
Time Frame: Week 56
Population: ITT set
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
percentage of participants | 30.14

19. Secondary Outcome: Percentage of Participants Who Were Week 8 Responders With Mucosal Healing at Week 8
Description: Mucosal healing was defined as an endoscopy sub-score of 0 or 1 at Week 8. Endoscopic findings were scored on a scale from 0 to 3 (higher score, worse disease): 0=Normal or inactive disease; 1=Mild disease (erythema, decreased vascular pattern, mild friability); 2=Moderate disease (marked erythema, lack of vascular pattern, friability, erosions); 3=Severe disease (spontaneous bleeding, ulceration). Clinical response was defined as reduction in complete full Mayo score of ≥ 3 points and ≥ 30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥ 1 point or absolute rectal bleeding subscore of ≤ 1 point at Week 8. Mayo score measures disease activity for ulcerative colitis from 0 (normal or inactive disease) to 12 (severe disease), calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and PGA), each ranging from 0 (normal) to 3 (severe disease). Negative change in Mayo score indicates improvement.
Time Frame: Week 8
Population: ITT set. A participant was a Week 8 responder if they had a clinical response at Week 8.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
percentage of participants | 39.04

20. Secondary Outcome: Percentage of Participants Who Were Week 8 Responders With Mucosal Healing at Week 56
Description: Mucosal healing was defined as an endoscopy sub-score of 0 or 1 at Week 56. Endoscopic findings were scored on a scale from 0 to 3 (higher score, worse disease): 0=Normal or inactive disease; 1=Mild disease (erythema, decreased vascular pattern, mild friability); 2=Moderate disease (marked erythema, lack of vascular pattern, friability, erosions); 3=Severe disease (spontaneous bleeding, ulceration). Clinical response was defined as reduction in complete full Mayo score of ≥ 3 points and ≥ 30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥ 1 point or absolute rectal bleeding subscore of ≤ 1 point at Week 8. Mayo score measures disease activity for ulcerative colitis from 0 (normal or inactive disease) to 12 (severe disease), calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and PGA), each ranging from 0 (normal) to 3 (severe disease). Negative change in Mayo score indicates improvement.
Time Frame: Week 56
Population: ITT set. A participant was a Week 8 responder if they had a clinical response at Week 8.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 76
percentage of participants | 46.05

21. Secondary Outcome: Change in Partial Mayo Score From Baseline to Week 8 in Participants Who Were Clinical Responders at Week 56
Description: The partial Mayo score is based on the Mayo score, which is a tool designed to measure disease activity for ulcerative colitis.
  The partial Mayo score (Mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding and PGA), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in partial Mayo score indicates improvement.
Time Frame: Baseline, Week 8
Population: ITT set of participants who were clinical responders at Week 56
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 55
score on a scale | 1.89 (1.61)

22. Secondary Outcome: Change in Full Mayo Score From Baseline to Week 8 in Participants Who Were Clinical Responders at Week 56
Description: Clinical response was defined as reduction in complete full Mayo score of ≥ 3 points and ≥ 30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥ 1 point or absolute rectal bleeding subscore of ≤ 1 point at Week 8. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and physician's global assessment [PGA]), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Baseline, Week 8
Population: ITT set of participants who were clinical responders at Week 56 with evaluable data for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 46
score on a scale | 3.17 (2.29)

23. Secondary Outcome: Change in Full Mayo Score From Baseline to Week 56 in Participants Who Were Clinical Responders at Week 56
Description: as for outcome 22
Time Frame: Baseline, Week 56
Population: ITT set of participants who were clinical responders at Week 56
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 55
score on a scale | 2.38 (2.06)

24. Secondary Outcome: Fecal Calprotectin Level at Week 8
Description: Fecal calprotectin is an indicator of inflammation in the colon with higher levels indicative of higher levels of inflammation.
Time Frame: Week 8
Population: ITT set.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
mg/kg | 456.89 (480.65)

25. Secondary Outcome: Fecal Calprotectin Level at Week 56
Description: as for outcome 24
Time Frame: Week 56
Population: ITT set.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Adalimumab
Number analyzed (Participants) | 146
mg/kg | 380.17 (466.93)

26. Secondary Outcome: Fecal Calprotectin Level at Week 8 in Participants Who Were Clinical Responders at Week 8
Description: as for outcome 24
Time Frame: Week 8
Population: ITT set. A participant was a Week 8 responder if they had a clinical response at Week 8 and had evaluable data for this outcome.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Adalimumab
Number analyzed (Participants) | 67
mg/kg | 336.33 (450.33)

27. Secondary Outcome: Fecal Calprotectin Level at Week 56 in Participants Who Were Clinical Responders at Week 8
Description: as for outcome 24
Time Frame: Week 56
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Adalimumab
Number analyzed (Participants) | 36
mg/kg | 281.87 (375.15)

28. Secondary Outcome: Fecal Calprotectin Level at Week 8 in Participants Who Were Clinical Responders at Week 56
Description: Fecal calprotectin is an indicator of inflammation in the colon with higher levels indicative of higher levels of inflammation. Clinical response was defined as reduction in complete full Mayo score of ≥3 points and ≥30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point at Week 8. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and PGA), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Week 8
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Adalimumab
Number analyzed (Participants) | 50
mg/kg | 464.58 (511.81)

29. Secondary Outcome: Fecal Calprotectin Level at Week 56 in Participants Who Were Clinical Responders at Week 56
Description: Fecal calprotectin is an indicator of inflammation in the colon with higher levels indicative of higher levels of inflammation. Clinical response was defined as reduction in complete full Mayo score of ≥3 points and ≥30% from Baseline (Week 0) with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point at Week 8. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and physician's global assessment [PGA]), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Week 56
Population: ITT set of participants who were clinical responders at Week 56 and had evaluable data for this outcome
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Adalimumab
Number analyzed (Participants) | 38
mg/kg | 415.40 (490.94)

30. Secondary Outcome: Change in the Composition of Fecal Microbiota From Baseline to Week 8 and Week 56
Description: Composition of fecal microbiota (16S ribosomal ribonucleic acid (rRNA) gene sequencing) was measured at Week 0, Week 8, and Week 56. Fecal bacterial composition was determined using 16S sequencing. The obtained sequences were analyzed using the Ezbiocloud database and 16S microbiome pipeline to assess composition and diversity.
Time Frame: Week 0, Week 8, Week 56
Population: This endpoint was not completed due to lack of data collection.
Arm/Group | Adalimumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Safety data were collected from the time of the participant's registration into the study until 70 days after study completion. Serious adverse events (SAEs) were reported to AbbVie from the time the physician obtained the participant's authorization to use and disclose information (or the participant's informed consent) until 70 days following the intake of the last dose of adalimumab taken during the study.
Description: As per the study protocol, all SAEs and adverse events (AEs) leading to adalimumab discontinuation were actively solicited. Any non-serious AEs were collected as spontaneous reports if AbbVie was notified. All SAEs and AEs leading to adalimumab discontinuation during this study period were reported to AbbVie regardless of their causal relationship to adalimumab.
Groups:
- Adalimumab: Adalimumab administered at 160 mg at week 0, 80 mg at week 2, and then 40 mg every other week per the Korean label.
Arm/Group | Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/146
Serious Adverse Events (participants affected / at risk) | 9/146
Other Adverse Events (participants affected / at risk) | 5/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=146)
Colitis ulcerative (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=146)
Haematochezia (Gastrointestinal disorders) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was an observational study in routine clinical practice. Inherent limitations leading to potential bias were lack of randomization and small number of intent to treat participants who completed the study without any major protocol deviations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/63/NCT02499263/SAP_000.pdf
  • Study Protocol (2016-09-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT02499263/Prot_001.pdf